CLINICAL TRIAL: NCT07129954
Title: Fear of Falling in Muscular Dystrophy: Investigation of the Phenomenon and a Multidisciplinary Rehabilitation Approach to Treat it
Brief Title: Fear of Falling in Muscular Dystrophy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universita di Verona (Other)
Responsible Party: Principal Investigator, Valentina Varalta, Doctor, Universita di Verona
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 561CET
Record Dates: First submitted 2025-08-11; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Fear of Falling; Duchenne Muscular Dystrophy (DMD); Muscular Dystrophies; Rehabilitation
Keywords: Fear of Falling; Muscular Dystrophy; Rehabilitation
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Muscular Dystrophies | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motor Rehabilitation (Active Comparator): Motor rehabilitation will be characterized by sessions of 45 minutes each with a patient (total sessions 36)
  Interventions: Behavioral: Motor rehabilitation
- Motor rehabilitation + cognitive behavioral therapy (Experimental): 1 session per week of 45 minutes of cognitive behavioral therapy and 2 sessions per week of 45 minutes of motor rehabilitation. The length of the treatment is the same as the control group: 12 weeks for 12 CBT sessions and 24 motor rehabilitation sessions (a total of 36 sessions).
  Interventions: Behavioral: Motor Rehabilitation and Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Motor rehabilitation — Motor rehabilitation will be characterized by sessions of 45 minutes each with a patient (total sessions 36): physiotherapist ratio of 1:1. The rehabilitation project will be defined by the PM&R specialist and the physiotherapist who will take charge of the patient. The treatment will focus on the maintenance of active and passive joint ranges, on the training of balance and gait, and on exercises of proprioception and scenic reinforcement. Specific devices (rehabilitation beds, verticalizer, posturography platform) will be used during motor treatment
  Arms: Motor Rehabilitation
Behavioral: Motor Rehabilitation and Cognitive Behavioral Therapy — 1 session per week of 45 minutes of cognitive behavioral therapy and 2 sessions per week of 45 minutes of motor rehabilitation. The length of the treatment is the same as the control group: 12 weeks for 12 CBT sessions and 24 motor rehabilitation sessions (a total of 36 sessions).
  Motor rehabilitation will be the same as that provided to the control group. In addition, participants will receive Cognitive-Behavioral Therapy (CBT), consisting of individual 45-minute sessions (one psychotherapist per patient).
  The sessions will focus on the relationship between cognition, emotions, and behavior. Specifically, the therapist will work with the patient to identify and modify automatic thoughts, cognitive distortions, and underlying beliefs or patterns associated with the fear of falling.
  Arms: Motor rehabilitation + cognitive behavioral therapy

SUMMARY:
Primary objectives

WP1: Evaluate the prevalence of FOF in the study population and how this varies over time. Evaluate whether there are relationships between the variables investigated (clinical, motor, cognitive, psychological) and the presence of FOF.

WP2: To evaluate, among those who presented disabling FOF, the effects of two different therapeutic approaches: motor rehabilitation vs. motor rehabilitation plus cognitive-behavioral psychotherapy.

Secondary objectives

WP1: To evaluate whether different profiles defined by specific clinical, motor, cognitive, psychological, and personological characteristics can be characterized among patients with dystrophy and FOF and how these impact functionality, activity, participation, and quality of life.

WP2: Evaluate the effects of cognitive-behavioral therapy (CBT) and a motor treatment on cognitive and psychological aspects, the frequency of falls, and the functional validity.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of muscular dystrophy: myotonic, facio-scapular-humeral, Becker, cingulate, Emery-Dreifuss, and distal;
* 16 to 65 years of age;
* Patients with residual walking capacity: functional ambulation category (FAC) at least equal to 1
* MMSE corrected for age and education of 23,8 points.

Specific Work Package 2 (WP2) inclusion criterion:

- the persistence of Fear Of Falling at 3 months, identified as a score of at least 16 points at the Falls efficacy scale - International (FES-I);

Exclusion Criteria:

* The presence of factors that may lead to the assumption that it is a priori impossible to ensure adequate adherence to the proposed treatment;
* Concurrent management in other rehabilitation centers or participation in other research projects
* Language barrier;
* Failure to sign informed consent.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-07-02 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Falls Efficacy Scale-International (FES-I) | The Falls Efficacy Scale - International (FES-I) will be administered at Baseline (T0), at 3 months (T1), at 6 months (T3), and at 9 months (T5).
  it allows us to identify the severity of the fear of falling. It consists of 16 questions directed to the patient, each of which can receive a score from 1 (=not at all concerned) to 4 (=very concerned). The scale range is from 16 to 64, where a lower score indicates less fear of falling. Specifically, a score between 16-19 indicates absent/mild fear of falling, between 20-27 moderate, and between 28-64 high (Morgan et al., 2013).

SECONDARY OUTCOMES:
North Star Ambulatory Assessment (NSAA) | it will be administered at 3 months (T1).
  to assess motor functionality. It is a scale consisting of 17 items that assess the performance of different functional skills, graded on a scale from 0 (unable), 1 (completed independently but with modifications), to 2 (completed without compensation. NSAA measures functional motor abilities in ambulant children with Duchenne Muscular Dystrophy (DMD). It is usually used to monitor the progression of the disease and treatment effects (Scott et al., 2012).
Posturographic examination | It will be administered at 3 months (T1), 6 months (T3), and 9 months (T5).
  to assess postural abilities. During the posturographic examinations, the amount of body oscillation is determined by recording the Centre of Pressure (COP) displacements over a period (Verbecque et al., 2016). Utilizing a posturographic platform for quantitative analysis offers enhanced accuracy and a deeper understanding of the patient's functional status. TYMO® device, a portable posturography platform, is employed to measure the tilts of the body's center of mass and track the outcomes of the rehabilitation process. This tool facilitates an objective, straightforward, and quantitative evaluation of the patient's functional status. The evaluative exercises offer various tests, including weight distribution assessment in force or percentage, balance assessment, equilibrium control assessment, and step counting.
Amount of walking | It will be measured one week before and one week after the rehabilitation intervention using a pedometer
  to assess walking functionality. The amount of walking will be measured one week before and one week after the rehabilitation intervention using a pedometer. To ensure maximum accuracy, participants will wear a watch all day except at night to track the number of steps.
Falls history | It will be collected at Baseline (T0).
  to assess the number of falls in the previous 3 months and any related consequences. During the first assessment, patients will be asked about the presence and number of falls in the last 3 months and the consequences of these falls.
Barthel index (BI) | It will be administered at Baseline (T0).
  to assess the level of disability. The Barthel Index, a scale used to assess the level of disability, consists of 10 items related to common daily activities (feeding, dressing/grooming, personal hygiene, bathing/showering, bladder continence, transferring from chair to bed, using the toilet, mobility/ambulation on level ground, climbing or descending stairs), investigating the degree of patient dependence/independence. The score for each item can be 0 (=dependent), 5 (=requires assistance), or 10 (=independent), with a maximum possible score of 100. A score below 100 indicates the presence of dependence (Mahoney et al.,1965).
Montreal Cognitive Assessment (MoCA) | It will be administered at 3 months (T1), 6 months (T3), and 9 months (T5).
  to assess cognitive global status. It is a screening tool for overall cognitive functioning consisting of 12 subtests exploring the following cognitive domains: memory (scores 0-5), visuospatial abilities (score 0-4), executive functions (score 0-4), attention, concentration, and working memory (score 0-6), language (score 0-6), spatial and temporal orientation (score 0-6). The total score ranges from 0 to 30, with higher scores indicating better cognitive functioning (Santangelo et al., 2015).
Trail Making Test (TMT) | It will be administered at 3 months (T1), 6 months (T3), and 9 months (T5).
  to assess psychomotor speed, attentional set-shifting, and visual-spatial search speed. It is composed of two parts. In Part A, which investigates selective attention, the participant must connect 25 circled numbers (distributed in a standardized random layout) in ascending order. In Part B, which investigates attentional set-shifting, the participant must alternately connect circled numbers from 1 to 13 and circled letters from A to N (e.g., 1-A-2-B-3-C). There is also a third index consisting of the difference between the scores obtained in Part A and Part B, indicating psychomotor and visual-spatial search speed. The faster and more accurate the patient is, the more their performance will be within the norm (Siciliano et al., 2019).
Modified Five-Point Test (MFPT) | It will be administered at 3 months (T1), 6 months (T3), and 9 months (T5).
  to assess visuospatial fluency by measuring the ability and speed to initiate a mental programming task and self-monitoring and visuospatial fluency. The result is based on the number of correct and unique drawings generated in 3 minutes (UDs) and the total number of drawings created according to a strategy (CSs) (Cattelani et al., 2011).
Beck Depression Inventory-II (BDI) | It will be administered at 3 months (T1), 6 months (T3), and 9 months (T5).
  to assess depressive symptoms. It is a self-administered instrument that assesses the severity of depression in adult subjects. It consists of 21 items and yields a total score; a higher score indicates greater depressive symptoms (range 0-63). The scale includes different cut-offs depending on the severity of the symptoms: 0-13 mild depression, 14-19 moderate depression, 20-28 moderate depression, 29-63 severe depression (Montano, Flebus, 2006).
State-Trait Anxiety Inventory (STAI) | It will be administered at 3 months (T1), 6 months (T3), and 9 months (T5).
  to assess anxiety symptoms. The questionnaire consists of 40 items to which the subject must respond in terms of perceived intensity on a Likert scale from 1 to 4 (higher scores indicating greater anxiety symptoms). The items are grouped into two scales. The first one investigates state anxiety, conceived as a particular experience of helplessness or insecurity in the face of perceived harm that can lead to worry or escape and avoidance. The second investigates trait anxiety, the tendency to perceive stressful situations as dangerous and threatening and to respond to various situations with varying intensity (Pedrabissi, Santinello, 1989).
The Big Five Observer (BFO) | It will be administered at 3 months (T1).
  to define personality traits. It is a sheet for observing and evaluating individual and organizational behaviors and social attitudes toward others. It can be used in any situation requiring hetero or self-assessment activities. The BFO is grounded in the theoretical framework of the psycholinguistic approach, using terms that are understandable even to non-psychologists. It consists of 40 pairs of opposite adjectives (8 for each Big Five: Extraversion-Introversion, Agreeableness-Disagreeableness, Conscientiousness-Negligence, Neuroticism-Emotional Stability, Openness-Closedness of Mind) selected from the Italian language vocabulary to be evaluated on a 7-point Likert scale (Caprara et al., 1994).
Short Form Health Survey questionnaire (SF-36) | It will be administered at 3 months (T1).
  to assess patient's quality of life. It is a popular instrument for evaluating Health-Related. The SF-36 measures eight scales: physical functioning (PF), role physical (RP), bodily pain (BP), general health (GH), vitality (VT), social functioning (SF), role emotional (RE), and mental health (MH). Component analyses showed two distinct concepts measured by the SF-36: a physical dimension, represented by the Physical Component Summary (PCS), and a mental dimension, represented by the Mental Component Summary (MCS). All scales contribute in different proportions to scoring PCS and MCS measures (Apolone & Mosconi, 1998).

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliera Universitaria Integrata Verona - UOC di Neuroriabilitazione, Verona, verona, Italy